CLINICAL TRIAL: NCT03203096
Title: Randomized, Double-blind, Placebo-controlled Intervention Study About the Effects of Magnesium Supplementation Using Nutritional Supplements on the Stress Parameters of Students Preparing for Examination
Brief Title: Magnesium Supplementation in Stress Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protina Pharmazeutische GmbH (Industry)
Collaborators: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StressMag2017
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Stress Physiology
Keywords: magnesium, stress, metabolomics, heart rate variability
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): identically tasting and looking Placebo
  Interventions: Dietary Supplement: Placebo
- Magnesium (Active Comparator): Supplementation with 400 mg Magnesium from Magnesium Citrate / Magnesium Oxide once daily
  Interventions: Dietary Supplement: Magnesium

INTERVENTIONS:
Dietary Supplement: Magnesium — Magnesium citrate / Magnesium oxide
  Arms: Magnesium
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine how a 6-week magnesium supplementation with 400 mg magnesium from magnesium citrate/magnesium oxide affects stress parameters in students in exam preparation.

DETAILED DESCRIPTION:
The examinations are carried out in 70 students in exam preparation (6 weeks before exam). The target parameters are determined in blood and 24h-urine. Blood sampling takes place at confinement, after 3 weeks and at the end of the study (week 6). In addition, heart rate variability is determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy students in exam preparation

Exclusion Criteria:

* pregnancy
* any chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
blood sampling | 6 weeks
  measurement of stress metabolites
24h-urine | 6 weeks
  measurement of stress metabolites
heart rate variability | 6 weeks
  measurement of heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Biomed Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No